CLINICAL TRIAL: NCT02910986
Title: Latinas LEarning About Density (LLEAD Study)
Brief Title: Behavioral and Psychological Impact of Returning Breast Density Results to Latinas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Mountain Park Health Center (Unknown); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 16-003707; R01MD009682 (NIH); MC1936 (Other: Mayo Clinic)
Record Dates: First submitted 2016-09-08; First posted 2016-09-22 (Estimated); Results first posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
Keywords: Mammography; Breast Density; Hispanic
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Usual Care (No Intervention): Breast density notification using standard language reporting for dense and non-dense breasts within the mammogram results notification letter
- Enhanced (Active Comparator): Usual Care plus a written educational brochure
  Interventions: Behavioral: Written educational brochure
- Interpersonal (Active Comparator): Usual Care plus Enhanced plus interaction with a promotora (lay health educator)
  Interventions: Behavioral: Written educational brochure; Behavioral: Promotora interaction

INTERVENTIONS:
Behavioral: Written educational brochure — Written educational brochure about breast density
  Arms: Enhanced; Interpersonal
Behavioral: Promotora interaction — Promotora education about breast density
  Arms: Interpersonal

SUMMARY:
This study will examine behavioral and psychological outcomes of breast density notification using a 3-group randomized design comparing usual written notification to two educationally enhanced approaches.

DETAILED DESCRIPTION:
This is a 3-group randomized clinical trial to compare usual care to two educationally enhanced approaches to breast density notification. Usual care involves sending written notification along with the mammogram report; all women will receive usual care. In addition, some women will receive written educational materials about breast density, with or without interaction with a promotora (culturally congruent health educator). Study outcomes include short and long term assessments of psychological (anxiety, knowledge) and behavioral (continued mammography screening, discussion with primary care provider) outcomes. The study also includes qualitative inquiry and a cost analysis.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Attending screening mammography at Mountain Park Health Center
* Speak English or Spanish

Exclusion Criteria:

* Male
* Current diagnosis of breast cancer

Ages: 40 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1386 (Actual)
Dates: Start 2016-10-27 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Celine M. Vachon, Ph.D., Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mountain Park Health Center, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ridgeway JL, Jenkins SM, Borah BJ, Suman VJ, Patel BK, Ghosh K, Rhodes DJ, Norman A, Ramos EP, Jewett M, Gonzalez CR, Hernandez V, Singh D, Sosa M, Radecki Breitkopf C, Vachon CM. Evaluating educational interventions to increase breast density awareness among Latinas: A randomized trial in a Federally Qualified Health Center. Cancer. 2022 Mar 1;128(5):1038-1047. doi: 10.1002/cncr.34017. Epub 2021 Dec 2. PMID 34855208
- [Result] Patel BK, Ridgeway JL, Jenkins S, Rhodes DJ, Ghosh K, Borah B, Suman V, Norman A, Leaver J, Jewett M, Hruska C, Gonzalez C, Singh D, Vachon CM, Breitkopf CR. Breast Density Knowledge and Awareness Among Latinas in a Low-Resource Setting. J Am Coll Radiol. 2022 Jan;19(1 Pt B):155-161. doi: 10.1016/j.jacr.2021.08.025. PMID 35033304
- [Result] Austin JD, Jenkins SM, Suman VJ, Raygoza JP, Ridgeway JL, Norman A, Gonzalez C, Hernandez V, Ghosh K, Patel BK, Vachon CM. Breast Cancer Risk Perceptions Among Underserved, Hispanic Women: Implications for Risk-Based Approaches to Screening. J Racial Ethn Health Disparities. 2025 Apr;12(2):1150-1158. doi: 10.1007/s40615-024-01949-7. Epub 2024 Feb 21. PMID 38383839
- [Derived] Ghosh K, Jenkins SM, Ridgeway JL, Austin JD, Borah BJ, Patel B, Rhodes DJ, Norman AD, Ramos EP, Jewett M, Gonzalez CR, Hernandez V, Singh D, Vachon CM, Suman VJ. A randomized trial to evaluate the impact of breast density notification on anxiety, breast cancer worry, and perceived risk among Latinas at a federally qualified health center : Breast density notification and anxiety, breast cancer worry, and perceived risk among Latinas. BMC Womens Health. 2025 Jun 2;25(1):274. doi: 10.1186/s12905-025-03818-9. PMID 40452038
- [Derived] Patel BK, Ridgeway JL, Ghosh K, Rhodes DJ, Borah B, Jenkins S, Suman VJ, Norman A, Jewett M, Singh D, Vachon CM, Radecki Breitkopf C. Behavioral and psychological impact of returning breast density results to Latinas: study protocol for a randomized clinical trial. Trials. 2019 Dec 18;20(1):744. doi: 10.1186/s13063-019-3939-6. PMID 31852492

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 10 patients who were found to be ineligible (n=2) or withdrew consent prior to randomization.
Period: Overall Study
Arm/Group | Usual Care | Enhanced | Interpersonal
Started | 460 | 456 | 461
Completed | 349 | 334 | 260
Not Completed | 111 | 122 | 201
Not completed — non-Latina | 14 | 13 | 12
Not completed — Failure to return T! survey | 72 | 84 | 72
Not completed — T1 Survey not 14-180 post education | 25 | 25 | 115
Not completed — Withdrew after randomization prior to start of intervention | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: These analyses included 943 Latinas who completed the T0 and T1 surveys per protocol.
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Enhanced | Interpersonal | Total
Number analyzed (Participants) | 349 | 334 | 260 | 943
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 47 [43 to 53] | 46 [43 to 53] | 47 [44 to 52] | 47 [43 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 349 | 334 | 260 | 943
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 349 | 334 | 260 | 943
  Not Hispanic or Latino | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 349 | 334 | 260 | 943
Region of Enrollment [Number; unit: participants]
  United States | 349 | 334 | 260 | 943

OUTCOME MEASURES:

1. Primary Outcome: Knowledge of Breast Density as a Masking Factor at First Follow-up
Description: Percentage of women who provided an incorrect response as to whether dense breasts impact the ability of a mammogram to correctly detect cancer at T0 but provided a correct response at T1
  Comparisons of the difference between the intervention groups in percentage of women who provided an incorrect response as to whether dense breasts impact the ability of a mammogram to correctly detect cancer at T0 but provided a correct response to the question at T1
Time Frame: Baseline (T0) to first follow-up (T1, 2 weeks to 180 days from education end)
Population: 943 participants who completed baseline and first follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced | Usual Care | Interpersonal
Number analyzed (Participants) | 334 | 349 | 260
Participants | 101 | 104 | 100
Statistical Analysis 1: Comparison: Enhanced vs Usual Care vs Interpersonal; The percentage with improved knowledge (defined as having an incorrect response at T0 and a correct response at T1) was compared between study groups with chi-square tests; Test type: Superiority; p > 0.05, Chi-squared

2. Primary Outcome: Anxiety Short Term (Baseline T0 to First Follow-up T1)
Description: The State-Trait Anxiety Inventory-State (STAI-S) s a 20-item self-report assessment. Items are answered on a 4-point Likert scale ranging from 1 (not at all) to 4 (very much so), with the total score ranging from 20 to 80, with higher scores indicating higher levels of anxiety symptoms. Anxiety was dichotomized as: normal (STAI score < 30) or moderate to severe (STAI score ≥ 30). The primary outcome was the percentage of participants who maintained or decreased to 'normal' anxiety levels at T1 from T0.
Time Frame: Change from baseline anxiety (T0) to T1: 2 weeks to 180 days after education end
Population: 516 Latina participants with complete follow-up over all three time points
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Enhanced | Interpersonal
Number analyzed (Participants) | 199 | 186 | 131
Participants
  Decreased or stayed normal | 99 | 88 | 70
  Increased or stayed moderate/severe | 100 | 98 | 61
Statistical Analysis 1: Comparison: Usual Care vs Enhanced vs Interpersonal; Test type: Superiority; p = 0.56, Chi-squared — The priori threshold for statistical significance was 0.05

3. Primary Outcome: BC Risk Assessment - Survey
Description: Percentage of women who provided incorrect response at baseline (T0) but a correct response at 14 to 180 days after completion of education to the question: 'Women who have dense breasts are at greater risk for getting breast cancer' (true, false, or I don't know).
  Comparisons of the difference in percentage of women who provided correct response to the single question: 'Women who have dense breasts are at greater risk for getting breast cancer' (true, false, or I don't know) between intervention groups.
Time Frame: T0 (baseline) to T1 (14 to 180 days after completion of education)
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced | Usual Care | Interpersonal
Number analyzed (Participants) | 334 | 349 | 260
Participants | 114 | 110 | 95
Statistical Analysis 1: Comparison: Enhanced vs Usual Care vs Interpersonal; Test type: Superiority; p > 0.05, Chi-squared — The priori threshold for statistical significance was 0.05
Statistical Analysis 2: Comparison: Enhanced vs Usual Care; Test type: Other; difference between EC and UC = 2.6, 98.3% CI 2-sided [-6.0 to 11.2]
Statistical Analysis 3: Comparison: Usual Care vs Interpersonal; Test type: Other; difference between INT and UC = 5.0, 98.3% CI 2-sided [-4.3 to 14.3]
Statistical Analysis 4: Comparison: Enhanced vs Interpersonal; Test type: Other; difference between INT and ENH = 2.4, 98.3% CI 2-sided [-7.0 to 11.9]

ADVERSE EVENTS:
Time Frame: Patients completed T1 surveys within 14-180 days from the end of study education and T2 surveys were completed within 275-545 days from the end of study education
Description: Changes in anxiety were addressed as a primary endpoint. There were no other specific survey questions addressing other potential adverse events.
Arm/Group | Usual Care | Enhanced | Interpersonal
All-Cause Mortality (participants affected / at risk) | 0/349 | 0/334 | 0/260
Serious Adverse Events (participants affected / at risk) | 0/349 | 0/334 | 0/260
Other Adverse Events (participants affected / at risk) | 0/349 | 0/334 | 0/260

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2022-08-12): https://cdn.clinicaltrials.gov/large-docs/86/NCT02910986/Prot_SAP_000.pdf
  • Informed Consent Form: English Consent (2019-07-18): https://cdn.clinicaltrials.gov/large-docs/86/NCT02910986/ICF_001.pdf
  • Informed Consent Form: Spanish Consent (2019-07-18): https://cdn.clinicaltrials.gov/large-docs/86/NCT02910986/ICF_002.pdf